CLINICAL TRIAL: NCT05490849
Title: 68Ga-HX01 PET in Healthy Volunteers and Malignant Tumors Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0799
Record Dates: First submitted 2022-07-20; First posted 2022-08-08 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Gallium-68

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-HX01 PET scanning (Experimental): Determine if 68Ga-HX01 PET is safe and effective method for imaging of malignant tumors
  Interventions: Drug: 68Ga-HX01

INTERVENTIONS:
Drug: 68Ga-HX01 — For pharmacokinetics, healthy volunteer underwent 68Ga-HX01 PET imaging. Blood samples were collected at 25 min, 55 min, and 115 min after imaging agent injection, and urine specimens were collected at 28 min, 58 min, and 118 min after injection to measure radioactivity in blood and urine. PET/MR scans were performed at 30-50 min, 60-80 min, and 120-140 min after injection to understand absorption, distribution, and metabolism.
  Cancer patients,
  1. Subjects should have 68Ga-HX01 and 18F-FDG PET scans two days apart.
  2. Blood tests, liver and kidney function, tumor markers (CA125, CA199, CEA, etc.), and other biochemical markers must be performed one week prior to and after imaging.
  3. Tumor biopsies or surgical specimens should be evaluated histopathologically and immunostained for biomarkers associated with angiogenesis.
  Other Names: gallium-68 (68Ga)-HX01

SUMMARY:
Angiogenesis is essential in tumor growth, proliferation, progression, and metastasis. Overexpression of aminopeptidase N (APN/CD13) and/or integrin αvβ3 in endothelial and tumor cells is an essential marker of tumor-associated angiogenesis. It is highly expressed in malignant tissues such as ovarian and pancreatic cancer but less expressed in normal tissues. Therefore, CD13 and αvβ3 are important targets for diagnosis and efficacy assessment in ovarian and pancreatic cancer. Single receptor targeting probes have many disadvantages, such as relatively low binding affinity, short tumor retention time, and low tumor uptake. RGD (Arg-Gly-Asp) and NGR (Asp-Gly-Arg) are recognized peptide sequences targeting CD13 or αvβ3. PET imaging with 68Ga-HX01, a radionuclide 68Ga labeled peptide isomer formed from RGD and NGR, can be helpful for targeted diagnosis and efficacy assessment of malignant tumors.

This project proposes to use 68Ga-HX01 PET imaging in the diagnosis and staging of malignant tumors, i.e., ovarian and pancreatic cancer, and to compare the diagnostic efficacy of 68Ga-HX01 with the pathology gold standard. And this study was conducted to compensate for the lack of value of 18F-FDG PET imaging for the diagnosis and staging of malignant tumors by comparing 68Ga-HX01 with the commonly used 18F-FDG PET imaging.

DETAILED DESCRIPTION:
Malignant tumors are a prevalent cause of death in human diseases that pose a grave threat to human health. The prognosis can be considerably improved by early diagnosis and therapy. Nevertheless, the pathophysiology of various types of tumors varies, and the diagnosis and treatment of tumors continue to provide challenges.

Angiogenesis is essential in tumor growth, proliferation, progression, and metastasis. Overexpression of aminopeptidase N (APN/CD13) and/or integrin αvβ3 in endothelial and tumor cells is an essential marker of tumor-associated angiogenesis. It is highly expressed in malignant tissues such as ovarian and pancreatic cancer but less expressed in normal tissues. Therefore, CD13 and αvβ3 are important targets for diagnosis and efficacy assessment in ovarian and pancreatic cancer. Single receptor targeting probes have many disadvantages, such as relatively low binding affinity, short tumor retention time, and low tumor uptake. RGD (Arg-Gly-Asp) and NGR (Asp-Gly-Arg) are recognized peptide sequences targeting CD13 or αvβ3. PET imaging with 68Ga-HX01, a radionuclide 68Ga labeled peptide isomer formed from RGD and NGR, can be helpful for targeted diagnosis and efficacy assessment of malignant tumors.

This project proposes to use 68Ga-HX01 PET imaging in the diagnosis and staging of malignant tumors, i.e., ovarian and pancreatic cancer, and to compare the diagnostic efficacy of 68Ga-HX01 with the pathology gold standard. And this study was conducted to compensate for the lack of value of 18F-FDG PET imaging for the diagnosis and staging of malignant tumors by comparing 68Ga-HX01 with the commonly used 18F-FDG PET imaging.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

1. fully understand and voluntarily sign the informed consent form
2. male or female, age 18-65 years
3. body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women; body mass index (BMI) within the range of 19.0 to 26.0 kg/m2 (including threshold values)
4. no history of chronic or severe disorders of the cardiovascular, liver, kidney, pulmonary, blood and lymphatic, endocrine, immunological, mental, neuromuscular, or gastrointestinal systems over the past three years; and good general health
5. no abnormalities in the evaluation of vital signs and physical exam
6. have no intention of having children, use effective contraception freely, and have no intention of donating sperm or eggs during the experiment and for six months following the trial's completion
7. be able to communicate effectively with the investigator and to comprehend and adhere to the study's criteria

Cancer patients:

1. The subject or his or her legal guardian may sign the informed consent form
2. a commitment to comply with the study guidelines and to to work with the investigator during the duration of the study
3. patients with clinically suspected or confirmed, but not tumor-related, ovarian cancer, pancreatic cancer, or other malignancies (supporting evidence includes serum relevant tumor markers, imaging data such as ultrasound, CT, MRI, and histological pathological examination) and in good general health
4. pathological results to be obtained by biopsy or surgical resection

Exclusion Criteria:

Healthy volunteers:

1. allergic body
2. acute diseases diagnosed before the study
3. have undergone surgery within 6 months prior to the trial would affect the absorption, distribution, metabolism, or excretion of the drug
4. have used any medication (including prescription drugs, over-the-counter drugs, herbal medicines) within 2 weeks prior to the study
5. pregnant and lactating women

Cancer patients:

1. patients or their legal guardian are unable or unwilling to sign the informed consent form
2. incapacity to collaborate in the complete implementation of the study
3. a history of cancer or oncologic treatment
4. acute systemic diseases and electrolyte disturbances
5. pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of 68Ga-HX01 by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | 1 year
  Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after injection of the imaging agent, and urine specimens were collected at 28 minutes, 58 minutes and 118 minutes after injection to measure the radioactivity in the blood samples and urine.
Adverse events collection | 1 year
  Adverse events after the injection and scanning of healthy volunteers and patients will be followed up and assessed.
Concentration of tumor markers (e.g., carcinoembryonic antigen, CA125, CA199) in participants' blood | 1 year
  Concentrations of blood tumor markers (e.g., CA125, CA199, CEA) measured on the date closest to the participant's examination will be collected. A higher blood tumor marker concentration means a higher threat or stage of tumor malignancy.
Count of red blood cells, white blood cells, hemoglobin and platelets; mean corpuscular volume (MCV), hematocrit | 1 year
  Count of red blood cells, white blood cells, hemoglobin and platelets; mean corpuscular volume (MCV), hematocrit measured on the date closest to the participant's examination will be collected. Abnormal changes (increase or decrease) in the above indicators may imply that the patient is threatened by the disease, which needs to be evaluated in conjunction with the patient's medical history and clinical manifestations.
Concentration of alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), albumin and total protein in participants' blood | 1 year
  Concentrations of blood alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase (ALP), albumin and total protein measured on the date closest to the participant's examination will be collected. Higher concentrations of the above indicators mean that the patient's liver function is more impaired.
Glomerular filtration rate (GFR) | 1 year
  This test is a measure of how well the kidneys are removing wastes and excess fluid from the blood. It is calculated from the serum creatinine level using age and gender. As kidney function decreases, the GFR level decreases.
Blood Urea Nitrogen (BUN) | 1 year
  As kidney function decreases, the BUN level rises.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhang X, Gai Y, Ye T, Fan L, Xiu L, Ruan W, Hu F, Chen J, Lan X. Head-to-head evaluation of [18F]FDG PET/CT and [68Ga]Ga-HX01 PET/MR in sarcoma patients. Eur J Nucl Med Mol Imaging. 2025 Jul;52(8):2898-2905. doi: 10.1007/s00259-025-07130-4. Epub 2025 Feb 20. PMID 39976700
- [Derived] Zhang X, Yang B, Qin C, Song X, Lv X, Zeng D, Gai Y, Lan X. Clinical Translation of a Dual-Integrin alphavbeta3- and CD13-Targeting PET Tracer. Clin Nucl Med. 2025 Apr 1;50(4):332-337. doi: 10.1097/RLU.0000000000005647. Epub 2025 Jan 20. PMID 39847870